CLINICAL TRIAL: NCT05829512
Title: Translation, Reliability, and Validity of Turkish Version of the Working Ability, Location, Intensity, Days of Pain, Dysmenorrhea (WaLIDD) Score
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 83116987-215
Record Dates: First submitted 2023-03-31; First posted 2023-04-25 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-04

CONDITIONS: Dysmenorrhea; Dysmenorrhea Primary
Keywords: Dysmenorrhea; Turkish version; Reliability; Validity; WaLIDD score
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients group: Individuals with dysmenorrhea
  Interventions: Other: Validity and reliability study

INTERVENTIONS:
Other: Validity and reliability study — Face-to-face questionnaire study

SUMMARY:
Currently, there is no agreement in the use of standard questionnaires with adequate validation and structuring measures to classify the severity of dysmenorrhea. This may explain the variability in prevalence, conditions associated with absenteeism (work, school, etc.), or errors in the diagnostic approach to patients with pelvic pain. The aim of this study is to conduct a cross-cultural adaptation study of the Turkish version of the working ability, location, intensity, days of pain, dysmenorrhea (WaLIDD) score, a tool designed to allow the identification of women with dysmenorrhea and those at high risk of obtaining medical clearance for the general population.

DETAILED DESCRIPTION:
Dysmenorrhea is the most common gynecological condition worldwide, affecting 90% of women of reproductive age. It is usually characterized by various symptoms such as pain, nausea, fatigue, depression, diarrhea, headache, insomnia, anxiety, weakness. According to the pathophysiology of dysmenorrhea, it can be classified as primary dysmenorrhea in which there is no organic disease or secondary dysmenorrhea due to an underlying pelvic abnormality. Primary dysmenorrhea presents with spasmodic, crampy menstrual pain and discomfort in the absence of pelvic pathology, while secondary dysmenorrhea is associated with a specific pelvic pathology such as endometriosis, adenomyosis, or uterine fibroids. Working ability, location, intensity, days of pain, dysmenorrhea (WaLIDD) score is an outcome scale designed as a scale type questionnaire (ability to work, location, intensity, days of pain, dysmenorrhea) integrating the features of score dysmenorrhea. This study will prove whether the Turkish version of the WaLIDD score is valid and reliable in evaluating women with dysmenorrhea. Statistical Package for Social Sciences (SPSS), version 22.0 computer package program for Windows will be used for statistical analysis. Statistical data will be expressed as mean±standard deviation (X±SD), median or percent (%). One-Sample Kolmogorov Smirnov test will be used to show the parametric or nonparametric distribution of the data. To determine the reliability of the WaLIDD score, test-retest and internal consistency analyzes will be performed at 7-day intervals. The test-retest value will be evaluated with the Intraclass Correlation Coefficient (ICC) and the internal consistency analysis will be evaluated with the Cronbach α value. The convergent validity of the WaLIDD score will be made using Pearson correlation analysis after calculating the total scores obtained from the Premenstrual Syndrome Impact Questionnaire, Pain Disability Index, and Big Five Inventory-10 questionnaires. Statistical significance value will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Menstrual pain that begins within a few months or within 2 years of menarche
* Pain that starts just before or at the beginning of menstruation,
* Pain in the lower abdomen and back, which may radiate to the inner thighs or both
* Pain, episodic and cramping pain, rarely lasting more than 72 hours,
* Pain similar to one menstrual cycle and additional symptoms such as nausea and vomiting, fatigue, headache, dizziness and sleep disturbances,
* Do not have any diagnosed chronic disease or a past or present psychological disorder,
* Able to speak, read and write Turkish.

Exclusion Criteria:

* Those with psychiatric and cognitive effects such as psychosis, bipolar disorder, eating disorder, moderate or severe depression or somatic symptom disorder,
* Those who participate in psychotherapy because of dysmenorrhea symptoms (currently or in the past), women in pregnancy and lactation,
* Having acute suicidal tendencies, gynecological diseases (hysterectomy, oophorectomy, gynecological cancer, polycystic ovary syndrome, endometriosis, infertility),
* Those who have used antidepressants, benzodiazepines/antipsychotics, oral contraceptives or hormones (e.g. thyroid hormones) in the last 3 months or have had a change in their use,
* With any neurological disorder,
* Can't speak, read or write Turkish.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with dysmenorrhea between the ages of 18-45
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
Working ability, location, intensity, days of pain, dysmenorrhea (WaLIDD) score | at first assessment
  Working ability, location, intensity, days of pain, dysmenorrhea (WaLIDD) score consists of 4 items. It was designed as a scale-type questionnaire integrating features of dysmenorrhea: 1) Number of anatomical pain locations (no part of the body, lower abdomen, lumbar region, lower extremities, inguinal region), 2) Wong-Baker pain rating (does not hurt, hurts a little, hurts a little more, hurts even more, hurts a lot, hurts a lot more), 3) Number of painful days in the menstrual period (0, 1-2, 3-4, ≥5), and 4) Frequency of pain that prevents performing activities (never, almost never, almost always, always). Each item has a score between 0 and 3. The total score ranges from 0 to 12 points. An increased score indicates a greater degree of dysmenorrhea.
Premenstrual Syndrome Impact Questionnaire | at first assessment
  The Premenstrual Coping Measure was developed to assess the ability of Australian women aged 18-49 to cope with premenstrual symptoms. Each item of the five-point Likert-type scale, which consists of 5 sub-dimensions, is scored between 1 and 5. No evaluation is made on the Premenstrual Coping Measure total score. As the score obtained from the sub-dimensions of the scale increases, the ability to cope with premenstrual symptoms also increases. The lowest score is 27, the highest score is 135. Increasing score indicates better coping ability. Turkish version, validity and reliability study of Premenstrual Coping Measure was conducted.
Pain Disability Index | at first assessment
  The Pain Disability Index is a self-administered, short and easy scale that measures the extent to which the pain secondary to ongoing discomfort affects the daily life of the individual and the level of disability developed due to this reason. The scale consists of seven questions. The individual is asked to rate the effects of pain on seven functional activities of daily living, consisting of family-home responsibilities, leisure time, occupation, social activity, sexual life, and self-care, by giving a score of 0 to 10 for all questions (0= not prevent, 5=moderate prevents, 10= I'am completely inadequate). The total score ranges from 0 to 70. 40 and above means a high level of disability. High scores indicate that the disability is severe. Turkish version, validity and reliability study is available.
Big Five Inventory-10 | at first assessment
  Big Five Inventory-10 has been brought to the literature as an alternative and short version of Big Five Inventory-44. The scale consists of 10 items and 5 sub-dimensions. The scale was evaluated with a 5- point Likert-type rating, as "Strongly Disagree", "Slightly Disagree", "Neither Agree nor Disagree", "Agree Slightly" and "Strongly Agree". The statements numbered 1-3-4-5-7 in the scale were reversed. The lowest score is 10, the highest score is 50. Increasing score and decreasing score according to sub-scales express better and worse personality traits. Turkish version, validity and reliability study of Big Five Inventory-10 was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Merkez, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Derived] Arikan H, Erol E. Working ability, Location, Intensity, Days of Pain, Dysmenorrhea (WaLIDD): cross-cultural adaptation, reliability, and validity of the Turkish version. BMC Womens Health. 2025 Mar 22;25(1):133. doi: 10.1186/s12905-025-03673-8. PMID 40121462